CLINICAL TRIAL: NCT03536559
Title: A Phase 2, Randomized, DB-PC, Parallel Group Study for the Treatment of Visual Pathway Deficits In Chronic Optic Neuropathy to Assess the Efficacy, Safety, Tolerability and Pharmacokinetics of CNM-Au8 For Remyelination In Multiple Sclerosis
Brief Title: Nanocrystalline Gold to Treat Remyelination Failure in Chronic Optic Neuropathy In Multiple Sclerosis
Acronym: VISIONARY-MS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19 related enrollment challenges.
Sponsor: Clene Nanomedicine (Industry)
Collaborators: Clene Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNMAu8.201
Record Dates: First submitted 2018-05-02; First posted 2018-05-24 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Optic Neuropathy; Optic; Neuritis, With Demyelination
Keywords: gold; nanocrystal; multifocal visual evoked potential; full field visual evoked potential; low contrast vision; low contrast letter acuity; remyelination; demyelination
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Optic Nerve Diseases; Neuritis; Demyelinating Diseases

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, parallel group, placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drug formulations will be identical in appearance (size, shape, volume, color) and smell. The packaging and labeling will be designed to maintain blinding to the Investigator's team and to patients. There are no visible differences between the active drug, and placebo dosing units
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 15mg CNM-Au8 (Experimental): 15mg suspension of clean-surfaced, faceted, gold nanocrystals in 60ml of sodium bicarbonate buffered water
  Interventions: Drug: CNM-Au8
- 30mg CNM-Au8 (Experimental): 30mg suspension of clean-surfaced, faceted, gold nanocrystals in 60ml of sodium bicarbonate buffered water
  Interventions: Drug: CNM-Au8
- Placebo (Placebo Comparator): The matched placebo to be used in this study will consist of water, sodium bicarbonate, and food coloring to match volume and color of the experimental treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNM-Au8 — CNM-Au8 is a dark red/purple-colored liquid formulation consisting of a stable suspension of faceted clean surfaced elemental gold nanocrystals in buffered deionized water with a concentration of up to 0.5 mg/mL of gold. The formulation is buffered by sodium bicarbonate present at a concentration of 0.546 mg/mL. There are no other excipients. The drug product is formulated to be taken orally and will be provided in single dose HDPE containers. The study doses vary by the concentration of gold nanocrystals per milliliter in a volume of 60 mL.
  Arms: 15mg CNM-Au8; 30mg CNM-Au8
Drug: Placebo — Placebo is liquid with identical color and taste
  Arms: Placebo

SUMMARY:
The objective of this trial is to assess the efficacy and safety of CNM-Au8 as a remyelinating treatment for vision-impairing MS lesions in participants who have chronic vision impairment as a result of Relapsing-Remitting Multiple Sclerosis. The primary endpoint is to assess the efficacy and safety of CNM-Au8 as a remyelinating therapy in patients with stable RMS. The secondary endpoint is Change in Functional Composite Responder Analysis Score from Baseline to Week 24.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, placebo-controlled study of the efficacy, safety, and pharmacokinetics of CNM-Au8 in stable RRMS patients who have Chronic Optic Neuropathy evidence by low contrast letter acuity deficits at Screening.

Patients will be screened over a 6-week period. Patients who meet the inclusion criteria and none of the exclusionary criteria will be enrolled into the clinical study.

All enrolled patients will have their visual baseline established in both eyes by functional, electrophysiological (at participating research sites), and morphological tests.

For each patient, the eye with the worst Baseline LCLA score will be considered as the affected eye. The other eye will be considered as the fellow eye. If both eyes have the same LCLA score at Baseline, then one eye will be randomly selected by the statistician to assess as the designated affected eye. Efficacy endpoints will be assessed in both the affected and the fellow eyes. Patients will be randomized to one of three groups: placebo, or one of two doses of CNM-Au8. All patients will receive their randomized investigational product (IP) dose daily over at least 24 consecutive weeks during the Fixed Duration Treatment Period. The study will also have a blinded Variable Duration Treatment Period for up to an additional 24-weeks (up to a 48-week maximum blinded duration) until the last-patient enrolled completes his/her Week 24 study visit per the study scheme in Figure 2. When the last enrolled patient completes his or her Week 24 visit, patients enrolled in the Variable Duration Treatment Period will complete the End-of-Study (EOS) visit at their next scheduled study visit.

The primary efficacy outcome measure will be assessed Efficacy will be assessed as an improvement in best-corrected low contrast letter acuity (BC-LCLA). Safety will be assessed up through the frequency of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and discontinuations due to adverse events (AEs), and changes in safety assessments (e.g., vitals, ECG, C-SSRS).

The study will remain blinded until the study database is locked.

All patients who are discontinued from treatment will complete the End-of-Study (EOS) assessment.

At the end of the Variable Duration Treatment Period, patients will complete an EOS assessment and then may choose either to exit the study, or receive open-label CNM-Au8 in a separate Open-Label Safety Extension Study.

An independent DSMB will be responsible for monitoring the safety of the study on a quarterly basis and ad hoc at the request of the DSMB or the Sponsor (e.g., in the event of unexpected SAEs) to review data throughout the Fixed Duration Treatment Period and the Variable Duration Treatment Period. The DSMB may make recommendations on the conduct of the study, including study termination. Appropriate procedures will be detailed in a DSMB Charter that will define disclosure of any findings along with patient- and study-stopping criteria.

There will be four study periods:

1. A six-week screening period (Screening Period);
2. A fixed 24-week double-blind, randomized treatment period (Fixed Duration Treatment Period);
3. A variable-duration, double-blind treatment period (Variable Duration Treatment Period) where patients continue the previously randomized treatment for up to an additional 24 weeks (total blinded duration of 48- weeks). This period will end for all patients when the last-enrolled patient reaches his or her 24-week visit (LP-24Wk) at which time patients in the Variable Duration Treatment Period will complete the EOS Visit at their next scheduled study visit;
4. A four-week follow-up period (Safety Follow-Up Period) for patients not continuing in the separate Open-Label Long-Term Safety Extension Study.

Following the end of the blinded treatment period, all patients who complete the 24-week Fixed Duration Treatment Period may be eligible to receive open-label CNM-Au8 in a separate Open-Label Long-Term Safety Extension Study.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and up to 55 years of age (inclusive) at Screening.
2. Clinical diagnosis of Relapsing Multiple Sclerosis (meeting McDonald criteria, 2010) who have had RMS no longer than 15 years from diagnosis.
3. Maximum Best Corrected High Contrast Visual Acuity (BC-HCVA) deficit on the Early Treatment Diabetic Retinopathy Study (ETDRS) Chart of 20/200 (6/60 metric) in both eyes.

   a. BC-HCVA is defined as the last line on the Early Treatment Diabetic Retinopathy Study (ETDRS) Chart that a patient is able to read three (3) or more letters correctly.
4. Best Corrected Low Contrast Letter Acuity (BC-LCLA) (by 2.5% Sloan Chart) must be 20/40 (6/12 metric) (inclusive) or worse in the affected eye and 20/32 (6/9.5 metric) or worse in the fellow eye; and the BC-LCLA must be worse than BC-HCVA for the respective value in both eyes.

   a. BC-LCLA is defined as the last line on the 2.5% Sloan Chart that a patient is able to read three (3) or more letters correctly.
5. Retinal Nerve Fiber Layer (RNFL) thickness ≥ 70 μm.
6. Stable disease activity based on the investigator's judgment over the previous 6 months.
7. All hematological parameters and biochemical parameters that fall outside the Within Normal Limits range must be assessed as Not Clinically Significant (NCS) and deemed stable or transient in nature.
8. Able to understand and give written informed consent.

Exclusion Criteria:

1. History of AQP4, MOG Ab(+) status, or ≥ 3 segments lesion in the spinal cord.
2. Any diagnosis other than RMS that could explain the patient's signs and symptoms.
3. An acute optic neuritis episode within the prior 6 months.
4. Clinical relapse requiring systemic steroid treatment within the prior 3 months (pre- treatment with systemic steroids during the administration of disease-modifying therapies [DMT] may be allowed after discussion with the Sponsor's Medical Monitor but must not be administered within 30 days of a planned VEP or MRI assessment).
5. Unstable treatment with a disease-modifying therapy (DMT) defined as a treatment change within prior 3-months unless due to intolerability.
6. Current treatment with immunosuppressive or immunomodulatory therapy other than those approved for the treatment of MS.
7. Any treatment with drugs known or suspected of producing retinal or optic nerve toxicity including hydroxychloroquine, chloroquine, clofazimine, vigabatrin, or ethambutol.
8. Any history of ophthalmological cause for retinal damage other than MS (e.g. cataracts, uveitis, macular degeneration, macular exudate, macular edema, glaucoma, severe astigmatism, ocular trauma, neuromyelitis optica, ischemic optic neuropathy, congenital nystagmus, retinal detachment, amblyopia, optic disk drusen).
9. Severe refractive defects: refractive errors (-6 dioptres to +6 dioptres or more in either eye, or axial eye length >26 mm), hypermetropia (> 6 dioptres; cylinder > 3 dioptres); or based on the investigators judgment any other ophthalmic diseases that would confound the study results or assessment of Visual Evoked Potential (VEPs), Best Corrected Visual Acuity (BCVA), Low Contrast Letter Acuity (LCLA), or Optical Coherence Tomography (OCT).
10. History diabetic retinopathy or a previous diagnosis of Diabetes Mellitus or history of prior impaired fasting glucose ≥126 mg/dL (or ≥ 200 mg/dL after oral glucose tolerance test).
11. History of human immunodeficiency virus (HIV), hepatitis C (HepC) virus antibody, or hepatitis B (HepB) virus antibody.
12. History of gold allergy.
13. Patients taking stimulant medications (including: amphetamine, dextroamphetamine, lisdexamfetamine, methylphenidate, or modafinil) who have not been on a stable dose greater than or equal to 30 days. Changes to dose will not be allowed during the course of the trial).
14. Patients taking clemastine fumarate, 4-aminopyridine (fampridine), or high dose Biotin (>300 mg/day).
15. Females who have a positive serum pregnancy test result at Screening or Baseline, or who are pregnant, breastfeeding, or planning to conceive during the study or within 180 days after study completion.
16. History or evidence of substance abuse or alcohol abuse within 5 years prior to Screening, including alcoholism; or severe tobacco use (>1 pack/day).
17. Clinical history of toxic neuropathy (e.g., secondary to treatment with ethambutol, isoniazid, linezolid, gentamycin, chloramphenicol, vincristine, or penicillamine).
18. Current enrollment in any other drug or device treatment study within 3 months prior to Baseline. Participation in an observational non-interventional study (i.e., no drug or device therapy) is not an exclusion criterion.
19. Inability to undergo any planned study procedures such as LCLA, VEP, MRI, or OCT; history of severe hypersensitivity to gadolinium-DTPA or reduced renal clearance (GFR must be ≥ 45 mL/min at Screening), claustrophobia; or inability to comply with study requirements based on Investigator judgment.
20. Patients with clinically significant hepatic or renal dysfunction or clinical laboratory findings that would limit the interpretability of change in liver or kidney function, or those with low platelet counts (< 150 x 10^9 per liter) or eosinophilia (absolute eosinophil count of ≥ 500 eosinophils per microliter) at Screening.
21. Based on the investigator's judgment, concurrent chronic or acute illness or unstable medical condition that may deteriorate that could confound the results of safety assessments, increase risk to the patient, or lead to difficulty complying with the protocol; including severe disc edema or hemorrhage, any clinically significant cardiac, endocrinological, hematological, hepatic, immunological, metabolic, urological, pulmonary, neurological (any progressive neurological disorder other than RRMS), dermatological, psychiatric (any untreated or unstable psychiatric disease including depression, bipolar and psychosis), renal, severe allergic or anaphylactic reactions, autoimmune, or other major confounding diseases.
22. Any history of previous malignancy, with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix, post documented full resections, with clean margins.
23. Patient is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Measures of Visual Function | Baseline to 48 weeks
  Change in Best-Corrected Low-Contrast Letter Acuity (BC-LCLA) score:
  Mean change in BC-LCLA from Baseline to Week 48 in the most affected eye as measured by 2.5% low contrast Sloan letter charts.

SECONDARY OUTCOMES:
Other Measures of Neurological Function | Baseline up to 48 weeks
  Change in the MS Functional Composite assessed by:
  Change from baseline for the average of the Z-scores of the six (m)MSFC domains.
  Combined ranked sum score for each (m)MSFC domain to the end of study. Time to the first repeated improvement of any two (m)MSFC domains by >=15%.

OTHER OUTCOMES:
Multifocal Visual Evoked Potential (mfVEP) Latency | Every 12 weeks following the 6-month primary endpoint, up to 48-weeks
  mfVEP latency is an electrophysiologic measure of remyelination that assesses the speed of conduction of electrical signals in neurons of the visual system.
Multifocal Visual Evoked Potential (mfVEP) Amplitude | Every 12 weeks following the 6-month primary endpoint, up to 48-weeks
  mfVEP amplitude is an electrophysiologic measure of axonal protection that assesses the magnitude of electrical signals in neurons of the visual system.
Full field Visual Evoked Potentials (ff-VEP) latency | At three month intervals beginning at 12-weeks, up to 48-weeks
  ffVEP latency is an electrophysiologic measure of remyelination that assesses the latency of electrical signals conduction in neurons of the visual system.
Full field Visual Evoked Potentials (ff-VEP) amplitude | At three month intervals beginning at 12-weeks, up to 48-weeks
  ffVEP amplitude is an electrophysiologic measure of axonal protection that assesses the magnitude of electrical signals in neurons of the visual system.
Optical Coherence Tomography (OCT) | At three month intervals beginning at 24-weeks, up to 48-weeks
  Measure of optic nerve morphology and retinal layers
Magnetic Resonance Imaging (MRI) | At three month intervals beginning at 24-weeks, up to 48-weeks
  Structural imaging of MS lesions
Change in Best High Contrast Visual Acuity Testing (HCVA) | Every 6-weeks, up to 48-weeks
  Mean change from Baseline in best-corrected high contrast visual acuity (BC-HCVA) score, as measured by EDTRS in the affected and fellow eye.
Expanded Disability Status Scale (EDSS) | At three month intervals beginning at 12-weeks, up to 48-weeks
  Standardized MS functional scales
9-Hole Peg Test | Every 12-weeks, up to 48-weeks
  Standardized test of upper body extremity function
Symbol Digit Modality Test (SDMT) | At three month intervals beginning at 12-weeks, up to 48-weeks
  Pattern matching functional scale
National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) | At three month intervals beginning at 12-weeks, up to 48-weeks
  Visual Function Quality of Life Scales
Ten-item Neuro-Ophthalmic Supplement (10-item NOS) | At three month intervals beginning at 12-weeks, up to 48-weeks
  Visual Function Quality of Life Scales
Six-Minute Walk Test (6MWT) | At three month intervals beginning at 12-weeks, up to 48-weeks
  Standardized Measure of Mobility and Exercise Tolerance
Timed 25-Foot Walk Test | Every 12-weeks, up to 48-weeks
  Quantitative mobility and leg function performance test
Individual OR Lesion MRI Analysis | Week 24 and week 48.
  Mean change in optic radiation lesional/non-lesional fibre DTI Divided by the MTR difference from Baseline.
Myelin Water Fraction MRI Analysis | Week 24 and Week 48
  Myelin Water Fraction (MWF) will be assessed with mcDESPOT imaging
Whole Brian Diffusion Tensor Imaging (DTI) divided by Magnetization Transfer Ratio (MTR) | Week 24 and week 48
  Mean change in whole brain DTI / MTR from Baseline.
Whole Brian White Matter Diffusion Tensor Imaging (DTI) divided by Magnetization Transfer Ratio (MTR) | Week 24 and week 48
  Mean change in whole brain white matter DTI / MTR from Baseline.
Whole Brian Lesion Diffusion Tensor Imaging (DTI) divided by Magnetization Transfer Ratio (MTR) | Week 24 and week 48
  Mean change in whole brain lesion DTI / MTR from Baseline.
Optic Radiation Diffusion Tensor Imaging (DTI) divided by Magnetization Transfer Ratio (MTR) | Week 24 and week 48
  Mean change in optic radiation DTI / MTR from Baseline.
Optic Radiation Lesion Diffusion Tensor Imaging (DTI) divided by Magnetization Transfer Ratio (MTR) | Week 24 and week 48
  Mean change in optic lesion radiation DTI / MTR from Baseline.
Change in Best Corrected Low-Contrast Letter Acuity (BC-LCLA) | Baseline up to 48 weeks
  Mean change by eye from Baseline in BC-LCLA score as determined by 2.5% low contrast Sloan letter chart for the affected and fellow eye. Proportion of patients with an improvement of at least 7 character letters by 2.5% low contrast Sloan letter chart in the affected and fellow eye.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Beadnall, MD, Principal Investigator — University of Sydney
Locations (7):
- UT Southwestern Medical Center, Dallas, Texas, United States
- Australia (5):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Sydney Brain Mind Centre, Sydney, New South Wales
  - Princess Alexandria Hospital, Woolloongabba, Queensland
  - Menzies Institute for Medical Research, Hobart, Tasmania
  - Alfred Health, Melbourne, Victoria
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No